CLINICAL TRIAL: NCT03758612
Title: A Phase 1, Partially-Blinded, Placebo-Controlled, Randomized, Single Ascending Dose (SAD) With a Food Effect Cohort Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TBI-223 in Healthy Adult Participants.
Brief Title: A Phase 1 Study to Evaluate Safety, Tolerability, and Pharmacokinetics of TBI-223 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TBI-223-CL-001
Record Dates: First submitted 2018-11-20; First posted 2018-11-29 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary
Keywords: TB; Tuberculosis; TBI-223; Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study is partially blinded. The repeat cohort (3b) using a different dosage formulation in Part 1 and subjects in Part 2 will be non-randomized and unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- TBI-223 50 mg (Active Comparator): Cohort 1, single dose of TBI-223 50 mg dosed under fasted conditions
  Interventions: Drug: TBI-223 oral suspension
- TBI-223 100 mg (Active Comparator): Cohort 2, single dose of TBI-223 100 mg dosed under fasted conditions
  Interventions: Drug: TBI-223 oral suspension
- TBI-223 300 mg (Active Comparator): Cohort 3a, Period 1 - gave a single dose of TBI-223 300 mg oral suspension dosed under fasted conditions.
  Cohort 3b, Period 2 - participants in cohort 3a were invited after a washout period to return for an additional single dose of TBI-223 300 mg enteric capsule dosed under fasted conditions
  Interventions: Drug: TBI-223 oral suspension; Drug: TBI-223 enteric capsule
- TBI-223 600 mg (Active Comparator): Cohort 4, single dose of TBI-223 600 mg dosed under fasted conditions
  Interventions: Drug: TBI-223 oral suspension
- TBI-223 1200 mg (Active Comparator): Cohort 5, Period 1, single dose of TBI-223 1200 mg dosed under fasted conditions.
  Cohort 5, Period 2, participants were invited to return after a washout period to continue in period 2 and receive a single dose of TBI-223 1200 mg dosed under fed conditions
  Interventions: Drug: TBI-223 oral suspension
- TBI-223 2000 mg (Active Comparator): Cohort 6, single dose of TBI-223 2000 mg dosed under fasted conditions
  Interventions: Drug: TBI-223 oral suspension
- TBI-223 2600 mg (Active Comparator): Cohort 7, single dose of TBI-223 2600 mg dosed under fasted conditions
  Interventions: Drug: TBI-223 oral suspension
- TBI-223 placebo (Placebo Comparator): Period 1 Single dose matching placebo for TBI-223 under fasted conditions for cohorts 1 to 7
  Period 2 Placebo participants in cohort 5 were invited to return after a washout period and were administered a single dose matching placebo for TBI-223 1200mg under fed conditions
  Interventions: Drug: Placebo suspension
- TBI-223 3x600 mg SR-1 tablet (Active Comparator): Cohort 8, arm 1 - Single dose TBI-223 of 1800 mg (3 x 600 mg) sustained release (SR) tablet formulation 1 under fed conditions
  Interventions: Drug: TBI-223 SR Tablet Prototype 1
- TBI-223 3x600 mg SR-2 tablet (Active Comparator): Cohort 8, arm 2 - Single dose TBI-223 of 1800 mg (3 x 600 mg) sustained release (SR) tablet formulation 2 under fed conditions
  Interventions: Drug: TBI-223 SR Tablet Prototype 2
- TBI-223 2x900 mg SR-3 tablet (Active Comparator): Cohort 8, arm 3 - Single dose TBI-223 of 1800 mg (2 x 900 mg) sustained release (SR) tablet formulation 3 under fed conditions
  Interventions: Drug: TBI-223 SR Tablet Prototype 3
- TBI-223 2x1000 mg IR tablet (Active Comparator): Cohort 8, arm 4 - Single dose TBI-223 of 2000 mg (2 x 1000 mg) immediate release (IR) tablet under fasted conditions
  Cohort 9 - Participants from cohort 8 arm 4 were invited to return and were administered a single dose TBI-223 of 2000 mg (2 x 1000 mg) immediate release (IR) tablet under fed conditions
  Interventions: Drug: TBI-223 IR Tablet

INTERVENTIONS:
Drug: TBI-223 oral suspension — TBI-223 oral suspension, orally administered.
  Arms: TBI-223 100 mg; TBI-223 1200 mg; TBI-223 2000 mg; TBI-223 2600 mg; TBI-223 300 mg; TBI-223 50 mg; TBI-223 600 mg
Drug: TBI-223 enteric capsule — TBI-223 enteric capsules filled with 150 mg of TBI-223 powder, orally administered.
  Arms: TBI-223 300 mg
Drug: TBI-223 SR Tablet Prototype 1 — TBI-223 600 mg sustained-release (SR) tablet Prototype 1, orally administered.
  Arms: TBI-223 3x600 mg SR-1 tablet
Drug: TBI-223 SR Tablet Prototype 2 — TBI-223 600 mg SR tablet Prototype 2, orally administered.
  Arms: TBI-223 3x600 mg SR-2 tablet
Drug: TBI-223 SR Tablet Prototype 3 — TBI-223 900 mg SR tablet Prototype 3, orally administered.
  Arms: TBI-223 2x900 mg SR-3 tablet
Drug: TBI-223 IR Tablet — TBI-223 1000 mg immediate release (IR) tablet, orally administered
  Arms: TBI-223 2x1000 mg IR tablet
Drug: Placebo suspension — Placebo for TBI-223 oral Suspension; orally administered.
  Arms: TBI-223 placebo

SUMMARY:
Partially-Blinded, Placebo-Controlled, Randomized, Single Ascending Dose (SAD) with a Food Effect Cohort to Evaluate the Safety, Tolerability, and Pharmacokinetics of TBI-223 in Healthy Adults.

DETAILED DESCRIPTION:
This study was a partially-blinded, placebo-controlled, randomized SAD study conducted at one study center. The primary objective of the study was to evaluate the safety and tolerability of single doses of TBI-223 oral suspension, TBI-223 oral enteric capsules, and TBI-223 tablet formulations in healthy adult subjects. The secondary objectives of the study were to determine the PK of TBI-223 and its metabolite M2 after single doses of TBI-223 oral suspension, TBI-223 oral enteric capsules, and TBI-223 tablet formulations in healthy adult subjects, and to compare the rate and extent of absorption of a single dose of TBI-223 oral suspension and TBI-223 tablet formulations when administered in healthy adult subjects either after a high-calorie, high-fat meal or in the fasting state.

Safety was assessed throughout the study for all subjects. Safety assessments included physical examinations, vital signs, serial ECGs, cardiac monitoring, adverse events (AEs), and clinical laboratory tests (including hematology, serum chemistry, coagulation, and urinalysis).

ELIGIBILITY:
Key Inclusion Criteria:

All volunteers must satisfy the following criteria to be considered for study participation:

1. Is a healthy adult male or female, 19 to 50 years of age (inclusive) at the time of screening.
2. Has a body mass index (BMI) ≥18.5 and ≤32.0 (kg/m2) and a body weight of no less than 50.0 kg.
3. Is medically healthy with no clinically significant screening results (e.g., laboratory profiles normal or up to Grade 1 per Division of Microbiology and Infectious Diseases Toxicity Tables), as deemed by the Investigator.
4. Has not used tobacco- or nicotine-containing products (including smoking cessation products), for a minimum of 6 months before dosing.
5. If assigned to receive study drug under fed conditions, is willing and able to consume the entire high-calorie, high-fat breakfast meal in the timeframe required.

Key Exclusion Criteria:

1. History or presence of clinically significant cardiovascular (heart murmur), pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
2. Any presence of musculoskeletal toxicity (severe tenderness with marked impairment of activity, or frank necrosis).
3. Has a positive test for hepatitis B surface antigen, hepatitis C antibody, or HIV at screening.
4. QTcF interval >450 msec for males or >470 msec for females at screening, Day -1, or Day 1 (predose), or history of prolonged QT syndrome. For the triplicate 12-lead ECGs taken at screening and on Day -1, the average QTcF interval of the three 12-lead ECG recordings were used to determine qualification.
5. Family history of long-QT syndrome or sudden death without a preceding diagnosis of a condition that was causative of sudden death (such as known coronary artery disease, congestive heart failure, or terminal cancer).
6. History of any of the following:

   * Serotonin syndrome
   * Seizures or seizure disorders, other than childhood febrile seizures
   * Brain surgery
   * History of head injury in the last 5 years
   * Any serious disorder of the nervous system particularly one that lowered the seizure threshold.
7. Lactose intolerant.
8. History of sensitivity or contraindication to use of linezolid, tedizolid, or any study investigational products

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Nedelman, Study Chair — Global Alliance for TB Drug Development
Locations (1):
- Worldwide Clinical Trials (WCT), San Antonio, Texas, United States

REFERENCES:
- [Derived] Lombardi A, Pappas F, Bruinenberg P, Nedelman J, Taneja R, Hickman D, Beumont M, Sun E. Pharmacokinetics, tolerability, and safety of TBI-223, a novel oxazolidinone, in healthy participants. Antimicrob Agents Chemother. 2025 Apr 2;69(4):e0154224. doi: 10.1128/aac.01542-24. Epub 2025 Mar 11. PMID 40067046

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort 3b, period 2, was added in protocol version 3.0. Some participants chose to return for period 2 and new participants were enrolled for period 2 of cohort 3b.
Groups:
- TBI-223 50 mg: Cohort 1, single dose of TBI-223 50 mg oral suspension dosed under fasted conditions.
- TBI-223 100 mg: Cohort 2, single dose of TBI-223 100 mg oral suspension dosed under fasted conditions.
- TBI-223 300 mg: Cohort 3a, Period 1 - gave a single dose of TBI-223 300 mg oral suspension dosed under fasted conditions.
  Cohort 3b, Period 2 - participants in cohort 3a were invited after a washout period to return for an additional single dose of TBI-223 300 mg as powder in enteric capsules dosed under fasted conditions
- TBI-223 600 mg: Cohort 4, single dose of TBI-223 600 mg oral suspension dosed under fasted conditions.
- TBI-223 1200 mg: Cohort 5, Period 1, single dose of TBI-223 1200 mg oral suspension dosed under fasted conditions.
  Cohort 5, Period 2, participants were invited to return after a washout period to continue in period 2 and receive a single dose of TBI-223 1200 mg oral suspension dosed under fed conditions.
- TBI-223 2000 mg: Cohort 6, single dose of TBI-223 2000 mg oral suspension dosed under fasted conditions.
- TBI-223 2600 mg: Cohort 7, single dose of TBI-223 2600 mg oral suspension dosed under fasted conditions.
- TBI-223 Placebo: Period 1 Single dose matching placebo for TBI-223 oral suspension under fasted conditions for cohorts 1 to 7
  Period 2 Placebo participants in cohort 5 were invited to return after a washout period and were administered a single dose matching placebo for TBI-223 1200mg oral suspension under fed conditions
- TBI-223 2x1000 mg IR Tablet: Cohort 8, arm 4 - Single dose TBI-223 of 2000 mg (2 x 1000 mg) immediate release (IR) tablet under fasted conditions
  Cohort 9 Participants from Cohort 8 arm 4 were invited to return and were administered a single dose TBI-223 of 2000 mg (2 x 1000 mg) immediate release (IR) tablet under fed conditions
Period: Period 1
Arm/Group | TBI-223 50 mg | TBI-223 100 mg | TBI-223 300 mg | TBI-223 600 mg | TBI-223 1200 mg | TBI-223 2000 mg | TBI-223 2600 mg | TBI-223 Placebo | TBI-223 3x600 mg SR-1 Tablet | TBI-223 3x600 mg SR-2 Tablet | TBI-223 2x900 mg SR-3 Tablet | TBI-223 2x1000 mg IR Tablet
Started | 6 | 6 | 6 | 6 | 8 | 6 | 8 | 14 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 8 | 6 | 8 | 14 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period
Arm/Group | TBI-223 50 mg | TBI-223 100 mg | TBI-223 300 mg | TBI-223 600 mg | TBI-223 1200 mg | TBI-223 2000 mg | TBI-223 2600 mg | TBI-223 Placebo | TBI-223 3x600 mg SR-1 Tablet | TBI-223 3x600 mg SR-2 Tablet | TBI-223 2x900 mg SR-3 Tablet | TBI-223 2x1000 mg IR Tablet
Started | 0 | 0 | 6 | 0 | 8 | 0 | 0 | 2 | 0 | 0 | 0 | 6
Completed | 0 | 0 | 4 | 0 | 8 | 0 | 0 | 2 | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | TBI-223 50 mg | TBI-223 100 mg | TBI-223 300 mg | TBI-223 600 mg | TBI-223 1200 mg | TBI-223 2000 mg | TBI-223 2600 mg | TBI-223 Placebo | TBI-223 3x600 mg SR-1 Tablet | TBI-223 3x600 mg SR-2 Tablet | TBI-223 2x900 mg SR-3 Tablet | TBI-223 2x1000 mg IR Tablet
Started | 0 | 0 | 6 (4 participants were returning participants from Cohort 3a and 2 participants were newly enrolled participants who received only the TBI-223 Oral Suspension in oral enteric capsules) | 0 | 8 | 0 | 0 | 2 (2 placebo participants in cohort 5 were invited to return and participate in period 2 with the other cohort 5 participants.) | 0 | 0 | 0 | 6
Completed | 0 | 0 | 6 | 0 | 7 | 0 | 0 | 2 | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants to whom a treatment was randomly assigned. Note that participants in cohort 3 were added for period 2 to replace participants who declined to return after period 1 and the baseline description contains all participants for cohort 3.
Groups:
- TBI-223 Placebo: Part 1 Single dose matching placebo for TBI-223 under fasted conditions
  Placebo suspension: Placebo for TBI-223 oral Suspension; orally administered
- TBI-223 300 mg: Cohort 3a, Period 1 - single dose of TBI-223 300 mg oral suspension dosed under fasted conditions
  Cohort 3b, Period 2 - participants in Cohort 3a were invited after a washout period to return for an additional single dose of TBI-223 300 mg as powder in enteric capsules dosed under fasted conditions
- TBI-223 1200 mg: Cohort 5, Period 1, single dose of TBI-223 1200 mg dosed under fasted conditions
  Cohort 5, Period 2, participants were invited to return after a washout period to continue in period 2 and receive a single dose of TBI-223 1200 mg oral suspension dosed under fed conditions.
  TBI-223 oral suspension: TBI-223 oral suspension, orally administered.
- TBI-223 3x600 mg SR-1 Tablet: Cohort 8, arm 1 -Single dose TBI-223 of 1800 mg (3 x 600 mg) sustained release (SR) tablet formulation 1 under fed conditions
  TBI-223 SR Tablet Prototype 1: TBI-223 600 mg sustained-release (SR) tablet Prototype 1, orally administered.
- TBI-223 3x600 mg SR-2 Tablet: Cohort 8, arm 2 -Single dose TBI-223 of 1800 mg (3 x 600 mg) sustained release (SR) tablet formulation 2 under fed conditions
  TBI-223 SR Tablet Prototype 2: TBI-223 600 mg SR tablet Prototype 2, orally administered.
- TBI-223 2x900 mg SR-3 Tablet: Cohort 8, arm 3 -Single dose TBI-223 of 1800 mg (2 x 900 mg) sustained release (SR) tablet formulation 3 under fed conditions
  TBI-223 SR Tablet Prototype 3: TBI-223 900 mg SR tablet Prototype 3, orally administered.
- TBI-223 2x1000 mg IR Tablet: Cohort 8, arm 4 -Single dose TBI-223 of 2000 mg (2 x 1000 mg) immediate release (IR) tablet under fasted conditions
  Cohort 9 - Participants from Cohort 8 arm 4 were invited to return and were administered a single dose TBI-223 of 2000 mg (2 x 1000 mg) immediate release (IR) tablet under fed conditions
  TBI-223 IR Tablet: TBI-223 1000 mg immediate release (IR) tablet, orally administered
- Total: Total of all reporting groups
Arm/Group | TBI-223 Placebo | TBI-223 50 mg | TBI-223 100 mg | TBI-223 300 mg | TBI-223 600 mg | TBI-223 1200 mg | TBI-223 2000 mg | TBI-223 2600 mg | TBI-223 3x600 mg SR-1 Tablet | TBI-223 3x600 mg SR-2 Tablet | TBI-223 2x900 mg SR-3 Tablet | TBI-223 2x1000 mg IR Tablet | Total
Number analyzed (Participants) | 14 | 6 | 6 | 8 | 6 | 8 | 6 | 8 | 6 | 6 | 6 | 6 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (10.73) | 34.5 (9.79) | 32.3 (3.93) | 30 (7.45) | 37.2 (9.11) | 32.6 (8.81) | 38.7 (8.48) | 32.8 (7.81) | 39.2 (8.30) | 30.7 (4.89) | 34.2 (9.13) | 33.3 (8.31) | 34.1 (8.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 6 | 4 | 5 | 2 | 5 | 4 | 4 | 4 | 1 | 42
  Male | 12 | 3 | 4 | 2 | 2 | 3 | 4 | 3 | 2 | 2 | 2 | 5 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 2 | 3 | 5 | 4 | 3 | 1 | 5 | 2 | 2 | 4 | 4 | 43
  Not Hispanic or Latino | 6 | 4 | 3 | 3 | 2 | 5 | 5 | 3 | 4 | 4 | 2 | 2 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 2 | 3 | 2 | 3 | 3 | 1 | 3 | 0 | 2 | 1 | 29
  White | 8 | 1 | 4 | 5 | 4 | 4 | 3 | 7 | 3 | 6 | 4 | 5 | 54
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 6 | 6 | 8 | 6 | 8 | 6 | 8 | 6 | 6 | 6 | 6 | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events
Description: A treatment-related adverse event (AE) is defined for this study as any AE classified as possibly, probably or certainly related to the study drug. Adverse events (AEs) for participants who received at least one dose of study treatment were collected from the signing of informed consent till the end of study visit. An Investigator reviewed each AE collected and assessed its relationship to drug treatment based on all available information at the time of the completion of the study.
Time Frame: Day 1 - Day 11
Population: All participants who received at least one dose of study treatment. Note: participants are divided here into analysis groups based on the drug and formulation taken and fed vs fasted status at dosing. This puts some participants into more than one analysis group based on the design of the study.
Measure: Count of Participants; unit: Participants
Groups:
- TBI-223 Placebo: Part 1 Single dose matching placebo for TBI-223 cohorts 1 to 7
  Placebo suspension: Placebo for TBI-223 oral Suspension; orally administered.
- TBI-223 300 mg Oral Suspension: Cohort 3a, single dose of TBI-223 300 mg oral suspension dosed under fasted conditions
  TBI-223 oral suspension: TBI-223 oral suspension, orally administered.
- TBI-223 300 mg Oral Enteric Capsules: Cohort 3b, single dose of TBI-223 300 mg as powder in enteric capsules dosed under fasted conditions
  TBI-223 capsule: TBI-223 enteric capsules filled with 150 mg of TBI-223 powder, orally administered.
- TBI-223 1200 mg Fasted: Cohort 5, Period 1, single dose of TBI-223 1200 mg dosed under fasted conditions
  TBI-223 oral suspension: TBI-223 oral suspension, orally administered.
- TBI-223 1200 mg Fed: Cohort 5, Period 2, single dose of TBI-223 1200 mg dosed under fed conditions
  TBI-223 oral suspension: TBI-223 oral suspension, orally administered.
- TBI-223 2x1000 mg IR Tablet Fasted: Cohort 8, arm 4 - Single dose TBI-223 of 2000 mg (2 x 1000 mg) immediate release (IR) tablet under fasted conditions
  TBI-223 IR Tablet: TBI-223 1000 mg immediate release (IR) tablet, orally administered
- TBI-223 2x1000 mg IR Tablet Fed: Cohort 9 - Single dose TBI-223 of 2000 mg (2 x 1000 mg) immediate release (IR) tablet under fed conditions
  TBI-223 IR Tablet: TBI-223 1000 mg immediate release (IR) tablet, orally administered
Arm/Group | TBI-223 Placebo | TBI-223 50 mg | TBI-223 100 mg | TBI-223 300 mg Oral Suspension | TBI-223 300 mg Oral Enteric Capsules | TBI-223 600 mg | TBI-223 1200 mg Fasted | TBI-223 1200 mg Fed | TBI-223 2000 mg | TBI-223 2600 mg | TBI-223 3x600 mg SR-1 Tablet | TBI-223 3x600 mg SR-2 Tablet | TBI-223 2x900 mg SR-3 Tablet | TBI-223 2x1000 mg IR Tablet Fasted | TBI-223 2x1000 mg IR Tablet Fed
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 8 | 7 | 6 | 8 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 1 | 0 | 0 | 3 | 2

2. Secondary Outcome: Area Under the Plasma Concentration-time- Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf)
Description: AUC0-inf will be calculated from plasma concentrations of TBI-223 AND M2 and calculated as AUC0-inf = AUC0-t + Clast/λz, where λz is the apparent terminal elimination rate constant calculated by linear regression of the terminal linear portion of the log concentration versus time curve
Time Frame: predose (0 hour) and at 0.5, 1.0, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 16, 20, 24, 30, 36, 42, 48, and 72 hours after administration of the investigational product
Population: Participants are divided into analysis groups based on the drug and formulation taken and fed vs fasted status at dosing. Some participants are in more than one analysis group based on the design of the study. Two subjects from Cohort 7 experienced emesis at 1.17 h and 1.37 h, respectively, after dosing. Data for these subjects were excluded from analyses of PK outcome measures. AUCs for SR-1, SR-2, and SR-3 were normalized to the 2000 mg dose.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TBI-223 50 mg | TBI-223 100 mg | TBI-223 300 mg Oral Suspension | TBI-223 300 mg Oral Enteric Capsules | TBI-223 600 mg | TBI-223 1200 mg Fasted | TBI-223 1200 mg Fed | TBI-223 2000 mg | TBI-223 2600 mg | TBI-223 3x600 mg SR-1 Tablet | TBI-223 3x600 mg SR-2 Tablet | TBI-223 2x900 mg SR-3 Tablet | TBI-223 2x1000 mg IR Tablet Fasted | TBI-223 2x1000 mg IR Tablet Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL
  TBI-223 | 1640 (344) | 2730 (628) | 10700 (2100) | 8690 (1690) | 25500 (9580) | 45000 (13800) | 47700 (14300) | 107000 (17800) | 127000 (37800) | 71300 (18800) | 69500 (16000) | 82600 (19400) | 86400 (21200) | 100000 (27300)
  M2 | 663 (106) | 1080 (178) | 4640 (881) | 4020 (511) | 8889 (2020) | 15900 (2660) | 15800 (2580) | 32900 (7340) | 36700 (4800) | 22700 (5350) | 22700 (4770) | 28400 (7240) | 25100 (3790) | 26000 (3540)

3. Secondary Outcome: AUC0-t
Description: AUC0-t will be calculated from plasma concentrations of TBI-223. Area under the plasma concentration-time curve from time-zero to the time of the last quantifiable concentration (Clast), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 2
Population: Two subjects from Cohort 7 experienced emesis at 1.17 h and 1.37 h, respectively, after dosing. Data for these subjects were excluded from analyses of PK outcome measures. AUCs for SR-1, SR-2, and SR-3 were normalized to the 2000 mg dose. Participants are divided into analysis groups based on the drug and formulation taken and fed vs fasted status at dosing. Some participants are in more than one analysis group based on the design of the study.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TBI-223 50 mg | TBI-223 100 mg | TBI-223 300 mg Oral Suspension | TBI-223 300 mg Oral Enteric Capsules | TBI-223 600 mg | TBI-223 1200 mg Fasted | TBI-223 1200 mg Fed | TBI-223 2000 mg | TBI-223 2600 mg | TBI-223 3x600 mg SR-1 Tablet | TBI-223 3x600 mg SR-2 Tablet | TBI-223 2x900 mg SR-3 Tablet | TBI-223 2x1000 mg IR Tablet Fasted | TBI-223 2x1000 mg IR Tablet Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL
  TBI-223 | 1620 (343) | 2730 (631) | 10700 (2090) | 8640 (1690) | 25500 (9560) | 45900 (13000) | 47600 (14300) | 107000 (17800) | 127000 (37700) | 71000 (18900) | 69400 (16000) | 82600 (19400) | 86300 (21200) | 100000 (27300)
  M2 | 633 (108) | 1050 (177) | 4610 (885) | 3980 (516) | 8850 (2020) | 16400 (2840) | 15800 (2590) | 32800 (7340) | 36600 (4790) | 22500 (5420) | 22600 (4770) | 28300 (7230) | 25100 (3800) | 26000 (3530)

4. Secondary Outcome: Maximum Plasma Concentration, Determined Directly From Individual Concentration-time- Data (Cmax)
Description: Cmax will be calculated from plasma concentrations of TBI-223. Cmax is calculated as the maximum plasma concentration, determined directly from individual concentration-time- data
Time Frame: as for outcome 2
Population: Participants are divided into analysis groups based on the drug and formulation taken and fed vs fasted status at dosing. Some participants are in more than one analysis group based on the design of the study. Two subjects from Cohort 7 experienced emesis at 1.17 h and 1.37 h, respectively, after dosing. Data for these subjects were excluded from analyses of PK outcome measures. Cmax for SR-1, SR-2, and SR-3 were normalized to the 2000 mg dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TBI-223 50 mg | TBI-223 100 mg | TBI-223 300 mg Oral Suspension | TBI-223 300 mg Oral Enteric Capsules | TBI-223 600 mg | TBI-223 1200 mg Fasted | TBI-223 1200 mg Fed | TBI-223 2000 mg | TBI-223 2600 mg | TBI-223 3x600 mg SR-1 Tablet | TBI-223 3x600 mg SR-2 Tablet | TBI-223 2x900 mg SR-3 Tablet | TBI-223 2x1000 mg IR Tablet Fasted | TBI-223 2x1000 mg IR Tablet Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL
  TBI-223 | 506 (156) | 811 (201) | 3090 (664) | 1360 (610) | 5800 (2400) | 8530 (1030) | 9150 (2740) | 14800 (2650) | 16200 (4640) | 7040 (2010) | 9580 (3390) | 8490 (1670) | 12800 (2320) | 19700 (5640)
  M2 | 109 (15.7) | 196 (31.3) | 897 (195) | 489 (137) | 1410 (397) | 2240 (345) | 2210 (399) | 3550 (871) | 3650 (772) | 1830 (557) | 2430 (657) | 2480 (499) | 2770 (499) | 3620 (847)

5. Secondary Outcome: Time of the Maximum Plasma Concentrations (Tmax)
Description: Tmax will be calculated from plasma concentrations of TBI-223.
Time Frame: as for outcome 2
Population: Participants are divided here into analysis groups based on the drug and formulation taken and fed vs fasted status at dosing. This puts some participants into more than one analysis group based on the design of the study. Two subjects from Cohort 7 experienced emesis at 1.17 h and 1.37 h, respectively, after dosing. Data for these subjects were excluded from analyses of PK outcome measures.
Measure: Median (Full Range); unit: hours
Arm/Group | TBI-223 50 mg | TBI-223 100 mg | TBI-223 300 mg Oral Suspension | TBI-223 300 mg Oral Enteric Capsules | TBI-223 600 mg | TBI-223 1200 mg Fasted | TBI-223 1200 mg Fed | TBI-223 2000 mg | TBI-223 2600 mg | TBI-223 3x600 mg SR-1 Tablet | TBI-223 3x600 mg SR-2 Tablet | TBI-223 2x900 mg SR-3 Tablet | TBI-223 2x1000 mg IR Tablet Fasted | TBI-223 2x1000 mg IR Tablet Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours
  TBI-223 | 1.0 [0.500 to 1.00] | 1.50 [1.00 to 2.00] | 1.37 [1.00 to 1.53] | 5.00 [3.00 to 16.0] | 1.75 [1.00 to 4.00] | 1.50 [1.00 to 3.02] | 1.50 [0.500 to 3.00] | 1.52 [1.00 to 3.05] | 2.25 [1.50 to 5.00] | 7.00 [6.00 to 16.0] | 6.50 [4.00 to 8.00] | 7.50 [5.00 to 20.0] | 2.00 [1.00 to 3.00] | 3.00 [1.00 to 4.00]
  M2 | 1.00 [0.500 to 3.00] | 1.50 [1.00 to 3.00] | 1.50 [1.50 to 3.00] | 5.50 [3.00 to 16.0] | 2.50 [1.00 to 4.00] | 3.00 [2.00 to 4.00] | 3.00 [2.00 to 4.00] | 3.50 [3.00 to 4.03] | 4.00 [3.00 to 5.00] | 7.50 [7.00 to 16.0] | 7.50 [4.00 to 8.00] | 8.00 [5.00 to 20.0] | 3.00 [3.00 to 4.00] | 3.00 [1.50 to 4.00]

6. Secondary Outcome: The Observed Terminal Elimination Half-life (t1/2)
Description: T1/2 will be calculated from plasma concentrations of TBI-223 and calculated as T½ = ln(2)/λz
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | TBI-223 50 mg | TBI-223 100 mg | TBI-223 300 mg Oral Suspension | TBI-223 300 mg Oral Enteric Capsules | TBI-223 600 mg | TBI-223 1200 mg Fasted | TBI-223 1200 mg Fed | TBI-223 2000 mg | TBI-223 2600 mg | TBI-223 3x600 mg SR-1 Tablet | TBI-223 3x600 mg SR-2 Tablet | TBI-223 2x900 mg SR-3 Tablet | TBI-223 2x1000 mg IR Tablet Fasted | TBI-223 2x1000 mg IR Tablet Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours
  TBI-223 | 2.19 (0.239) | 1.96 (0.165) | 1.94 (0.238) | 3.43 (1.02) | 2.63 (0.693) | 2.93 (0.706) | 2.32 (0.158) | 3.81 (0.870) | 2.93 (0.534) | 3.70 (0.271) | 2.32 (0.581) | 3.08 (0.784) | 2.80 (0.604) | 2.38 (0.101)
  M2 | 2.62 (0.256) | 2.41 (0.238) | 2.25 (0.403) | 3.93 (1.36) | 3.17 (0.585) | 3.33 (0.635) | 2.72 (0.207) | 4.44 (0.698) | 3.74 (0.752) | 4.21 (2.45) | 2.77 (0.728) | 3.61 (0.843) | 3.24 (0.604) | 2.97 (0.325)

7. Secondary Outcome: Geometric Mean Ratio and 90% Confidence Interval (CI) of Cmax, AUC0-t and AUC 0-inf of 300 mg TBI-223 in Capsule to Oral Suspension Formulations
Description: Geometric mean ratio of TBI-223 area under the (plasma concentration vs. time) curve and Cmax when administered as a Single 300 mg Dose of TBI-223 Capsule Formulation (Cohort 3 Repeat; Part 1; Test) and a Single 300 mg Dose of TBI-223 Oral Suspension (Cohort 3; Part 1; Reference).
Time Frame: as for outcome 2
Population: Participants enrolled in cohort 3a and cohort 3b who received TBI-223. Participants from cohort 3a were invited to participate in cohort 3b and additional participants were enrolled in 3b to replace those who elected not to participate.
Measure: Geometric Mean (90% Confidence Interval); unit: ratio (%)
Groups:
- TBI-223 Ratio (%): Ratio(%) = Geometric Mean (Test)/Geometric Mean (Reference)
Arm/Group | TBI-223 Ratio (%)
Number analyzed (Participants) | 8
ratio (%)
  Cmax | 42.46 [31.57 to 57.10]
  AUC0-t | 94.43 [90.28 to 98.76]
  AUC0-inf | 94.73 [90.58 to 99.06]

8. Secondary Outcome: Geometric Mean Ratio and 90% Confidence Interval (CI) of Cmax, AUC0-t and AUC 0-inf of 1200 mg Oral Suspension Under Fasted to Fed Conditions
Description: Geometric mean ratio of TBI-223 area under the (plasma concentration vs. time) curve and Cmax when administered as a Single 1200 mg Dose of TBI-223 Oral Suspension under Fed (Test) and Fasted (Reference) Conditions (Part 1; Cohort 5)
Time Frame: as for outcome 2
Population: All participants who enrolled in cohort 5 and received TBI-223. Participants in period 1 were invited to participate in period 2.
Measure: Geometric Mean (90% Confidence Interval); unit: ratio (%)
Arm/Group | TBI-223 Ratio (%)
Number analyzed (Participants) | 8
ratio (%)
  Cmax | 103.34 [87.00 to 122.75]
  AUC0-t | 103.23 [97.80 to 108.96]
  AUC0-inf | 102.79 [96.37 to 109.64]

9. Secondary Outcome: Geometric Mean Ratio and 90% Confidence Interval (CI) of Cmax, AUC0-t and AUC 0-inf of 2000 mg of Immediate Release (IR) Tablets Under Fed to Fasted Conditions.
Description: Geometric mean ratio of TBI-223 area under the (plasma concentration vs. time) curve and Cmax when administered as IR tablets, 2000 mg (2 x 1000 mg TBI-223 tablets) under Fed Conditions (Cohort 9; Test) and IR tablets, 2000 mg (2 x1000 mg TBI-223 tablets) under Fasted Conditions (Cohort 8; Reference)
Time Frame: as for outcome 2
Population: All participants who enrolled were enrolled in cohort 8, arm 4 and were also enrolled in cohort 9.
Measure: Geometric Mean (90% Confidence Interval); unit: ratio (%)
Arm/Group | TBI-223 Ratio (%)
Number analyzed (Participants) | 6
ratio (%)
  Cmax | 151.24 [127.91 to 178.82]
  AUC0-t | 115.73 [112.08 to 119.50]
  ACU0-inf | 115.70 [112.06 to 119.47]

10. Secondary Outcome: Geometric Mean Ratio and 90% Confidence Interval (CI) of Cmax, AUC0-t and AUC 0-inf of TBI-223 1800 mg Sustained Release (SR) Tablets Under Fed Conditions to 2000 mg IR Tablets Under Fasted Conditions
Description: Geometric mean ratio of TBI-223 area under the (plasma concentration vs. time) curve and Cmax when administered as SR (Prototypes 1, 2, and 3) under Fed Conditions (Cohort 8; Test) and IR, 2000 mg (2 x 1000 mg TBI-223 tablets) under Fasted Conditions (Cohort 8; Reference)
Time Frame: as for outcome 2
Population: SR-1, SR-2, and SR-3 parameters were dose-normalized to 2000 mg prior to analysis
Measure: Geometric Mean (90% Confidence Interval); unit: ratio (%)
Groups:
- TBI-223 Ratio (%), SR-1 Fed vs IR Fasted; TBI-223 Ratio (%), SR-2 Fed vs IR Fasted; TBI-223 Ratio (%), SR-3 Fed vs IR Fasted: Ratio(%) = Geometric Mean (Test)/Geometric Mean (Reference)
Arm/Group | TBI-223 Ratio (%), SR-1 Fed vs IR Fasted | TBI-223 Ratio (%), SR-2 Fed vs IR Fasted | TBI-223 Ratio (%), SR-3 Fed vs IR Fasted
Number analyzed (Participants) | 12 | 12 | 12
ratio (%)
  Cmax | 53.53 [40.10 to 71.45] | 71.70 [53.71 to 95.71] | 66.31 [49.67 to 88.53]
  AUC0-t | 81.11 [62.92 to 104.56] | 80.55 [62.49 to 103.84] | 95.71 [74.25 to 123.38]
  AUC 0-inf | 81.52 [63.26 to 105.04] | 80.56 [62.51 to 103.81] | 95.73 [74.29 to 123.35]

11. Secondary Outcome: Geometric Mean Ratio and 90% Confidence Interval (CI) of Cmax, AUC0-t and AUC 0-inf of 1800 mg SR Tablets (Prototypes 1, 2, 3,) to 2000 mg IR Tablets Under Fed Conditions
Description: Geometric mean ratio of TBI-223 area under the (plasma concentration vs. time) curve and Cmax when administered as TBI-223 after 1800 mg SR tablets (Prototypes 1, 2, 3,) under Fed Conditions (Cohort 8; Test) and 2000 mg IR tablets (2 x 1000 mg TBI-223 tablets) under Fed Conditions (Cohort 8; Reference)
Time Frame: as for outcome 2
Population: SR-1, SR-2, and SR-3 parameters were dose-normalized to 2000 mg prior to analysis
Measure: Geometric Mean (90% Confidence Interval); unit: ratio (%)
Groups:
- TBI-223 Ratio (%), SR-1 Fed vs IR Fed; TBI-223 Ratio (%), SR-2 Fed vs IR Fed; TBI-223 Ratio (%), SR-3 Fed vs IR Fed: Ratio(%) = Geometric Mean (Test)/Geometric Mean (Reference)
Arm/Group | TBI-223 Ratio (%), SR-1 Fed vs IR Fed | TBI-223 Ratio (%), SR-2 Fed vs IR Fed | TBI-223 Ratio (%), SR-3 Fed vs IR Fed
Number analyzed (Participants) | 12 | 12 | 12
ratio (%)
  Cmax | 35.39 [26.04 to 48.10] | 47.41 [34.88 to 64.43] | 43.85 [32.26 to 59.59]
  AUC0-t | 70.09 [54.10 to 90.81] | 69.60 [53.72 to 90.18] | 82.70 [63.83 to 107.15]
  AUC0-inf | 70.45 [54.40 to 91.24] | 69.62 [53.76 to 90.17] | 82.74 [63.88 to 107.15]

ADVERSE EVENTS:
Time Frame: Day 1 - Day 11
Description: Subjects were instructed to inform the research personnel of any AEs that occurred at any time during the study. Subjects were monitored for AEs from the first dose through the end-of-study visit. Reported or observed AEs were documented and followed to resolution. Participants are divided here into analysis groups based on the drug and formulation taken and fed vs fasted status at dosing. This puts some participants into more than one analysis group based on the design of the study.
Groups:
- TBI-223 Placebo: Part 1 Single dose matching placebo for TBI-223
  Placebo suspension: Placebo for TBI-223 oral Suspension; orally administered.
- TBI-223 2x1000 mg IR Tablet Fasted: Cohort 8, arm 4 -Single dose TBI-223 of 2000 mg (2 x 1000 mg) immediate release (IR) tablet under fasted conditions
  TBI-223 IR Tablet: TBI-223 1000 mg immediate release (IR) tablet, orally administered
Arm/Group | TBI-223 Placebo | TBI-223 50 mg | TBI-223 100 mg | TBI-223 300 mg Oral Suspension | TBI-223 300 mg Oral Enteric Capsules | TBI-223 600 mg | TBI-223 1200 mg Fasted | TBI-223 1200 mg Fed | TBI-223 2000 mg | TBI-223 2600 mg | TBI-223 3x600 mg SR-1 Tablet | TBI-223 3x600 mg SR-2 Tablet | TBI-223 2x900 mg SR-3 Tablet | TBI-223 2x1000 mg IR Tablet Fasted | TBI-223 2x1000 mg IR Tablet Fed
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/7 | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/7 | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/14 | 1/6 | 2/6 | 1/6 | 0/6 | 0/6 | 0/8 | 1/7 | 3/6 | 3/8 | 1/6 | 2/6 | 2/6 | 3/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TBI-223 Placebo (N=14) | TBI-223 50 mg (N=6) | TBI-223 100 mg (N=6) | TBI-223 300 mg Oral Suspension (N=6) | TBI-223 300 mg Oral Enteric Capsules (N=6) | TBI-223 600 mg (N=6) | TBI-223 1200 mg Fasted (N=8) | TBI-223 1200 mg Fed (N=7) | TBI-223 2000 mg (N=6) | TBI-223 2600 mg (N=8) | TBI-223 3x600 mg SR-1 Tablet (N=6) | TBI-223 3x600 mg SR-2 Tablet (N=6) | TBI-223 2x900 mg SR-3 Tablet (N=6) | TBI-223 2x1000 mg IR Tablet Fasted (N=6) | TBI-223 2x1000 mg IR Tablet Fed (N=6)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Energy Increased (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT03758612/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT03758612/SAP_001.pdf